CLINICAL TRIAL: NCT05241951
Title: Preventing Medication-Related Problems in Care Transitions to Skilled Nursing Facilities Using a Pharmacy Integrated Transitional Team
Brief Title: Preventing Medication-Related Problems in Care Transitions to Skilled Nursing Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Giana Davidson, Associate Professor, School of Medicine: Surgery, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00011018; 1R01HS027805 (AHRQ)
Record Dates: First submitted 2022-01-28; First posted 2022-02-16 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Care Transition
Keywords: Care Transition; Medication-Related Problems; Post-Acute Care; Skilled Nursing Facility; Hospital Systems; Medication Safety
MeSH Terms: interventions — Remote Consultation

STUDY DESIGN:
Intervention Model Description: A parallel cluster-randomized controlled crossover trial design, with randomization occurring at the skilled nursing facility cluster level. The trial is conducted across four hospitals and 14 independent SNFs in Washington State. SNF's are stratified by patient volume before randomly assigned to either the PIT program or usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Pharmacist in Transition of Care (Experimental): A clinical pharmacist will be provided as a patient discharges from one of four University of Washington (UW) medical centers to one of 14 post acute skilled nursing facilities randomized to the intervention arm. The coordinating transitional pharmacist will conduct (1) a comprehensive medication review including medication reconciliation, adjustment, and monitoring during the transitional period from hospital to SNF, 2) a structured handoff between clinical teams at the hospital and SNF.
  Interventions: Other: Structured hand-off; Other: Medication reconciliation during transitional period; Other: Transitional medication monitoring; Other: Teleconsultation
- Patient transitions from hospital to post-acute care (No Intervention): Patient will transition from one of four University of Washington (UW) medical centers to one of 14 post-acute skilled nursing facilities randomized to the control arm. Patients will receive the standard discharge process.

INTERVENTIONS:
Other: Structured hand-off — Use of standardized checklist to provide synchronous or asynchronous handoff that conveys medication recommendations to the SNF clinical teams
  Other Names: Standardized Checklist
  Arms: Clinical Pharmacist in Transition of Care
Other: Medication reconciliation during transitional period — Comprehensive medication reconciliation conducted during transitional period between hospital and SNF, focused on SNF-specific requirements for medication delivery (e.g., stop dates, titration instructions)
  Arms: Clinical Pharmacist in Transition of Care
Other: Transitional medication monitoring — Review of medication orders during first 7 days of SNF admittance to address barriers to translation of medication orders and appropriate medication delivery
  Arms: Clinical Pharmacist in Transition of Care
Other: Teleconsultation — Ad hoc consultation to provide additional clarification to SNF clinical teams
  Arms: Clinical Pharmacist in Transition of Care

SUMMARY:
The Pharmacy Integrated Transitions (PIT) program, utilizes a crossover randomized control design to evaluate the impact of a clinical pharmacist in decreasing medication related problems during a patient's transition from hospital to skilled nursing facility (SNF).

DETAILED DESCRIPTION:
Standard hospital discharge processes (e.g. as recommended by the Joint Commission Center for Transforming Healthcare), include hospital staff completing a paper-based discharge summary and medication reconciliation form. To reduce the likelihood of medication-related problems during care transitions, the Pharmacy Integrated Transitions (PIT) program aims to improve the standard transition process by adding a coordinating transitional pharmacist to provide a structured synchronous "warm-handoff" between clinical teams at the hospital and the Skilled Nursing Facility, in addition to reconciling, adjusting, and monitoring medications during and after discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* patients receiving inpatient care at University of Washington Mountlake, University of Washington Northwest, Harborview, and Valley Medical Center hospitals to one of 14 collaborating SNF's on a day when the PIT program pharmacist is conducting the intervention

Exclusion Criteria:

* Under 18 years of age
* patients with a discharge on hospice care
* patients discharged on days that the pharmacist is not conducting the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1052 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Medication Related Problems | 30 days post hospital discharge
  Number of medication related problems experienced by patients within 30 days post hospital discharge.

SECONDARY OUTCOMES:
Death | 30 Days post hospital discharge
  Number of deaths experienced by patients within each cohort
Readmissions | 30 Days
  Number of readmissions within 30 days of index hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Giana Davidson, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Health System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers

REFERENCES:
- [Derived] Hantouli MN, Monsell SE, Davidson GH, Chaing J, Comstock B, Dervish AA, Gionet NJ, Howard S, Jimenez N, Kim C, Liberman M, Lindo EG, Marcum ZA, Ong TD, Serrano E, Simons K, Sun LS, Zaslavsky O, Austin E; PIT Collaborative. Pharmacy Integrated Transitions (PIT) trial: a protocol for a pragmatic cluster-randomised crossover trial. BMJ Open. 2024 Dec 31;14(12):e088786. doi: 10.1136/bmjopen-2024-088786. PMID 39740951
- See also: Focused on evaluating the effectiveness and value of healthcare and keeping the patient's voice central, CERTAIN is a revolutionary approach to improving quality through actionable research. — http://www.becertain.org/